CLINICAL TRIAL: NCT02511275
Title: Assessment of Nephrotoxicity Associated to Parenchymal Clamping During Partial Nephrectomy Using a Microdialysis Technique: NECPAR Study
Brief Title: Nephrotoxicity Associated to Parenchymal Clamping During Partial Nephrectomy Using a Microdialysis Technique
Acronym: NECPAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: this type of surgery is now performed with a surgical robot that no longer allows the realization of microdialysis
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: University Hospital of Saint-Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1308142; 2014-A00098-39 (Other: ANSM)
Record Dates: First submitted 2015-02-20; First posted 2015-07-30 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Nephrectomy; Kidney Cancer; Microdialysis
Keywords: parenchymal clamping; microdialysis technique; partial nephrectomy
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- renal microdialysis (Other): patient with renal microdialysis
  Interventions: Procedure: Renal microdialysis

INTERVENTIONS:
Procedure: Renal microdialysis — Renal microdialysis is an innovative and promising technique in the monitoring of renal ischemia. Its sterile nature enables intraoperative use to give us real-time reflection of the in situ metabolism. In Patients who participated in clinical research with this microinvasive technique, no complications including bleeding has been reported.

SUMMARY:
Surgery plays a central role in kidney cancer management being the only therapy that offers the possibility of healing the patients. Currently, the partial nephrectomy is a standard technique because it meets the principle of nephron sparing surgery. A partial nephrectomy requires a control of the renal blood flow using a clamp, which can be parenchymal or vascular (pedicular). In France, most of the centers use pedicular clamping. It is well established that this technique results in warm ischemia of the entire healthy parenchyma and can lead to permanent kidney damages. Currently, no study evaluated the impact of parenchymal clamping on the healthy parenchyma.

The aim of the investigators study is to evaluate the nephrotoxicity of the healthy parenchyma due to parenchymal clamping during partial nephrectomy. This assessment will be done through a microdialysis technique. The microdialysis probe is directly implanted in the healthy unclamped parenchyma and will allow us to measure in real time, during the surgery, the biological changes related to anaerobic metabolism of renal interstitial space. All those measures will be completed by urinary and plasmatic assessments. Oxidative stress will be assessed using four markers of tubular viability : Interleukin 18 (IL18), Kidney Injury Molecule-1 (KIM-1), Neutrophil Gelatinase-Associated Lipocalin (NGAL) and cystatin C and four parameters of anaerobic metabolism : lactate, pyruvate, glycerol and glucose.

This is a prospective pilot study limited to 10 patients included over 12 months. Depending on the results, it will be further developed by a second study comparing parenchymal with pedicle clamping.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the urological surgery department with an indication of partial nephrectomy
* Patients with a renal lesion classified T1 (≤7cm) or for T2 eligible to a partial nephrectomy and having an possibility to benefit from a parenchymal clamping (decided on preoperative imaging)

Exclusion Criteria:

* Patient with a chronic kidney disease (functional or structural renal abnormality evolving for more than three months and Glomerular Filtration Rate <60 ml/min)
* Patient carrying a renal lesion classified T1 but too close to the renal pedicle or not accessible for a parenchymal clamping
* Patients in whom tumor removal requires ice cooling or kidney pedicular clamping

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2015-03-10 (Actual); Study Completion 2015-03-30 (Actual)

PRIMARY OUTCOMES:
Average interstitial lactate concentrations (peak lactate and lactate/pyruvate ratio) | every 10 minutes unitl the end of clamping

SECONDARY OUTCOMES:
Interstitial concentrations of lactate, pyruvate, lactate/pyruvate ratio, glycerol concentration (marker of impaired cellular membrane) and glucose concentration | every 10 minutes until the end of clamping then every 300 minutes until the third hour of no-clamping
  composite measure
Blood and urine concentration of Interleukin 18 (IL18), le Kidney Injury Molecule-1 (KIM-1), le Neutrophil Gelatinase-Associated Lipocalin (NGAL) and Cystatin C | 1 hour before clamping, then Hour +2, Hour +6, Hour +12, Hour +24, Hour +36 ; Hour 0 corresponding to the timing of clamping
  composite measure
Preoperative creatinine | inclusion day and at 2 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MOTTET, MD PhD, Principal Investigator — CHU de Saint Etienne
Locations (1):
- Chu de Saint Etienne, Saint-Etienne, France